CLINICAL TRIAL: NCT06744478
Title: Assessing the Magnitude of Anisometropia in Patients Wearing Misight 1 Day Contact Lens
Status: Enrolling by invitation | Type: Observational
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB113-170-A
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Myopia; Anisometropia
MeSH Terms: conditions — Myopia; Anisometropia | interventions — Contact Lenses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- myopic children: Myopic children use Misight 1 Day Contact Lens every day for myopia and anisometropia control.
  Interventions: Device: Misight 1 Day Contact Lens

INTERVENTIONS:
Device: Misight 1 Day Contact Lens — Misight 1 Day Contact Lens wearing for myopia control

SUMMARY:
The effectiveness of Misight 1 Day Contact Lens in retarding anisometropic progression has not been investigated before. This study is aimed to elucidate the efficacy of Misight 1 Day Contact Lens for anisometropia control.

ELIGIBILITY:
Inclusion Criteria:

* 8-23 years old children diagnosed with anisometropia and are willing to accept MiSight® 1 Day contact lens wearing treatment.
* No congenital eye diseases or eye diseases such as strabismus and amblyopia.
* Those who have been stated to be willing to participate in the program for at least 24 months and accept various evaluations.

Exclusion Criteria:

* Ocular surface disease( dry eye, keratoconus..)
* Allergy to contact lens
* Received eye surgery before
* The cornea is infected (bacterial, fungal or viral infection).
* Strabismus
* Premature birth

Ages: 8 Years to 23 Years | Sex: All
Age Groups: Child, Adult
Study Population: We enroll the clinical patients who was diagnosed with anisometropia (meaning that myopia exceeds 100 degree diopters during the refraction examination, and the difference between the other eye is more than 100 degree diopters). Age limit was 8 to 23 years old. The purpose and process were carefully addressed to the subjects and their guardians who signed an informed consent form before commencing this study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of the visual acuity in myopic children with different Misight 1 Day Contact Lens | From the date of starting treatment, the visual acuity was measured 1 week, 1month and every 3 months up to 24 months.
  The investigators measure the visual acuity of myopic children with different Misight 1 Day Contact Lens.

SECONDARY OUTCOMES:
Changes of axial length in myopic children with different Misight 1 Day Contact Lens | From the date of starting treatment, the axial length was measured, then repeat measure were performed every 6 months up to 24 months
  The investigators measure the axial length(mm) of eyeball of myopic children with different diopter of Misight 1 Day Contact Lens.

CONTACTS AND LOCATIONS:
Locations (1):
- Shang-Yen WU, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided